## Statistical Analysis Plan

As far as we know there is no previous data on diaphragmatic disfunction incidence in the cohort group in study. The aim of the study is to provide an estimation of this disfunction incidence. There are about 30 estimated patients per year that may respond to inclusion and exclusion criteria in our hospital, so that us allow to calculate a 95% confidence interval (CI), with a maximal amplitude equal to 35.8%. The valuation of CI in relation to incidence is shown in the following table.

| Incidence % | CI 95% | | Total interval amplitude |
|-------------|--------|------|--------------------------|
| 10 | 0 | 20.7 | 20.7 |
| 20 | 5.7 | 34.3 | 28.6 |
| 30 | 13.6 | 46.4 | 32.8 |
| 40 | 22.5 | 57.5 | 35.1 |
| 50 | 32.1 | 67.9 | 35.8 |
| 60 | 42.5 | 77.5 | 35.1 |
| 70 | 53.6 | 86.4 | 32.8 |
| 80 | 65.7 | 94.3 | 28.6 |
| 90 | 79.3 | 100 | 20.7 |

## Data analysis

The frequence of diaphragmatic thickening fraction will be reported as a percentage with 95% relative CI in different time spans. Categorial variables will be described as absolute frequencies while continuous variables will be described with statistical average and standard deviation or median and interquartile range.